CLINICAL TRIAL: NCT04842006
Title: Systemic Neoadjuvant and Adjuvant Control by Precision Medicine in Rectal Cancer (SYNCOPE) - Approach on High-risk Group to Reduce Metastases
Brief Title: Systemic Neoadjuvant and Adjuvant Control by Precision Medicine in Rectal Cancer
Acronym: SYNCOPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Toni Seppala, Principal Investigator, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUS/155/2021
Record Dates: First submitted 2021-02-08; First posted 2021-04-12 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TNT + precision (Experimental)
  Interventions: Drug: Total neoadjuvant therapy (TNT); Diagnostic Test: Minimal residual disease (MRD)
- Conventional (Active Comparator)
  Interventions: Radiation: Long radiation therapy

INTERVENTIONS:
Drug: Total neoadjuvant therapy (TNT) — Short radiotherapy (5X5 Gy) and capecitabine/oxaliplatin
  Arms: TNT + precision
Diagnostic Test: Minimal residual disease (MRD) — Postoperative MRD on circulating cell-free DNA
  Arms: TNT + precision
Radiation: Long radiation therapy — Long-course 50.4 Gy radiation with capecitabine
  Arms: Conventional

SUMMARY:
Rectal cancer represents the most complex area of multidisciplinary treatment in bowel surgery. In 2017, there were 1221 new rectal cancers in Finland. The prognosis of colorectal cancer (CRC) patients these days is almost exclusively driven by the occurrence of the metastatic form of the disease.

The treatment of rectal cancer often includes a long delay between diagnosis and the initiation of systemic chemotherapy, increasing risk for systemic metastases for those at high risk. On the other hand, the waiting time during pretreatment before surgery enables comprehensive systematic characterization of the primary tumor status before the decisions on adjuvant chemotherapy, opening a window to the use of precision in decision-making.

In this randomized controlled treatment trial, outcomes of novel precision methods to select right rectal cancer patients for treatment that they need will be compared to conventional treatment. The study aims to reduce over-treatment of those that most likely do not benefit from additional treatments. With the overall aim to reduce metastatic form of the disease, patients with high-risk features will be randomized to a treatment strategy with early systemic control by chemotherapy followed by circulating tumor DNA (ctDNA) and organoid-guided adjuvant therapy, or to conventional treatment strategy. Both state-of-the-art laboratory practice and routine diagnostic clinical pipelines are introduced to bring future diagnostic models of minimal residual disease and chemoresistance closer to current practice. The outcomes will reveal the clinical benefit of such strategy by recurrence-free survival at highest level of evidence, and produce important clinical outcome data on the application of ctDNA in everyday cancer treatment practice. The translational data on the use of ctDNA organoids to inform treatment decision and regimen selection will build knowledge of the use of such biomarkers as tools for clinical practice and clinical research. The results will be scalable worldwide in the practice of rectal cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

1. rectal adenocarcinoma,
2. World Health Organization (WHO) performance status 0-1, assessed by the MDT to be able to undergo capecitabine and oxaliplatin (CAPOX) treatment, 3) extramural vein invasion by magnetic resonance imaging (mrEMVI+) and

4) assessed by the multi-disciplinary team (MDT) to require either radiotherapy (RT) or long chemoradiotherapy (CRT) by the current standards.

Exclusion Criteria:

1. deficient mismatch repair (MMR) status,
2. non-dihydropyrimidine dehydrogenase (DPYD) genotype,
3. a contraindication to capecitabine, oxaliplatin or RT, or
4. failing in blood tests that describe the adequate circulatory, liver and kidney function for chemotherapy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 3 years from surgery
Recurrence-free survival | 5 years from surgery
Postoperative ctDNA | 3 weeks postoperatively
  number of patients with detectable ctDNA at postoperative sample in the conventional treatment arm that are not assigned to chemotherapy

SECONDARY OUTCOMES:
CRC-specific survival | 3 years
CRC-specific survival | 5 years
overall survival | 3 years
overall survival | 5 years
number of surgically resected patients resected patients | 1 year
R0-resection rate | 1 year
local recurrence rate | 5 years postoperatively
complete pathological response response rate | 12 weeks after initiation of pretreatment
complete clinical response rate | 12 weeks after initiation of pretreatment
total uptake of chemotherapy | 1year
total uptake of chemotherapy | 3 years
total uptake of chemotherapy | 5 years
adverse effects of surgery effects of surgery | 1 year
adverse effects of chemotherapy | 1 year
adverse effects of chemotherapy | 3 years
Treatment response by patient-derived organoid (PDO) therapy response | 1 year
  population distribution of PDO treatment response is compared to their corresponding clinical response by response MRI and pathological response and compared to organoid in vitro response

CONTACTS AND LOCATIONS:
Overall Officials: Toni T Seppala, MD, PhD, Principal Investigator — Tampere University Hospital
Locations (2):
- Finland (2):
  - Helsinki University Central Hospital, Helsinki, Uusimaa
  - Tampere University Hospital, Tampere

IPD SHARING:
Plan to Share IPD: No